CLINICAL TRIAL: NCT03438461
Title: A Randomized, Open-label, Single-dose, 6-Period, 8-Sequence Crossover Study to Evaluate the Relative Oral Bioavailability of Seltorexant (JNJ-42847922) After Administration of 3 Different Formulations in Healthy Subjects Under Fasted and Semi-fasted Conditions
Brief Title: A Study to Evaluate the Relative Oral Bioavailability of Seltorexant (JNJ-42847922) After Administration of 3 Different Formulations in Healthy Participants Under Fasted and Semi-fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108446; 42847922MDD1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-02-08; First posted 2018-02-19 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — seltorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): In Part 1, all participants will receive a single oral dose of seltorexant (40 milligram [mg]) in all the 6 treatments as Treatment A (Formulation 1 in fasted state), B (Formulation 1 in semi-fasted state), C (Formulation 2 in fasted state), D (Formulation 2 in semi-fasted state), E (Formulation 3 in fasted state) and F (Formulation 3 in semi-fasted state) and the participants will be assigned to one of the 8 sequences (that is, ADBCEF, ADBCFE, BACDEF, BACDFE, CBDAEF, CBDAFE, DCABEF, DCABFE). A washout period of at least 7 days between subsequent study drug administrations on Day 1 of each treatment period will be maintained.
  Interventions: Drug: Seltorexant 40 mg
- Part 2 (Optional) (Experimental): Optional Part 2 will only be performed if considered to be warranted by the sponsor based on the preliminary pharmacokinetic (PK) analysis of the results from Part 1. Participants will receive a single oral dose of seltorexant (20 mg) as 3 different formulations assigned to one of the either 6 or 4 treatment sequences under fasted or semi-fasted conditions. The treatment will be assigned in 1 of the 6 or 4 assigned sequences per treatment period that is either Period 1 to 6 or Period 1 to 4).
  Interventions: Drug: Seltorexant 20 mg

INTERVENTIONS:
Drug: Seltorexant 40 mg — Seltorexant 40 mg as two tablets of 20 mg will be administered as Formulation 1, 2 and 3 orally in Part 1.
  Arms: Part 1
Drug: Seltorexant 20 mg — Seltorexant as a tablet of 20 mg will be administered as Formulation 1, 2 and 3 orally in Part 2.
  Arms: Part 2 (Optional)

SUMMARY:
The purpose of this study is to assess and compare the pharmacokinetics (PK) and relative oral bioavailability of 3 oral tablet formulations of seltorexant in fasted and semi-fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an informed consent form (ICF) indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* Willing to adhere to the prohibitions and restrictions specified in the study protocol
* If a woman of childbearing potential, must have a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test at screening and a negative urine pregnancy test on Day -1 of the first treatment period
* If a woman, must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 30 days after the last study drug administration
* A man, who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator (example, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Has a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic (Child-Pugh Score greater than or equal to [>=] 7) or renal insufficiency (estimated glomerular filtration rate [eGFR] less than (<) 60 milliliter per minute per 1.73 meter square (mL/min/1.73m^2) based on the modified diet renal disease [MDRD] formula determined at screening, thyroid disease, neurologic (including seizure disorders) or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results. Significant gastrointestinal past history, or any disease/surgery (excluding cholecystectomy and appendectomy) that would interfere with drug absorption
* Has clinically significant abnormal values for hematology, serum chemistry (including thyroid stimulating hormone [TSH] at screening only) or urinalysis at screening or at admission to the study site. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to both the investigator and to the Janssen Research & Development Safety Physician, are acceptable
* Has clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at screening or at admission to the study site as deemed appropriate by the investigator
* Has used any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol (acetaminophen), oral contraceptives, and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled or has used any systemic herbal medications or dietary supplements including products containing Hypericum perforatum (example, St. John's Wort) from 21 days before the first dose of study drug is scheduled
* Received a known inhibitor of CYP(cytochrome P450)3A4 or CYP2C9 activity within 14 days or a period less than 5 times the drugs half-life; whichever is longer, before the first dose of the study drug is scheduled

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) when Compared for 3 Oral Tablet Formulations of Seltorexant | Predose, 20 minutes (min), 30min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 20h (Day 1), 24h, 36h (Day 2), 48h (Day 3) postdose
  Cmax is the maximum observed plasma concentration and will be evaluated when compared for 3 oral tablet formulations of seltorexant in fasted and semi-fasted conditions.
Area Under the Plasma Concentration-Time Curve from the Time of Study Drug Administration to the Last Measurable Plasma Concentration (AUC[0-last]) when Compared for 3 Oral Tablet Formulations of Seltorexant | Predose, 20 minutes (min), 30min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 20h (Day 1), 24h, 36h (Day 2), 48h (Day 3) postdose
  AUC (0-last) is the area under the plasma concentration-time curve from the time of study drug administration to the last measurable plasma concentration and will be evaluated when compared for 3 oral tablet formulations of seltorexant in fasted and semi-fasted conditions.
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinite Time (AUC[0-infinity]) when Compared for 3 Oral Tablet Formulations of Seltorexant | Predose, 20 minutes (min), 30min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 20h (Day 1), 24h, 36h (Day 2), 48h (Day 3) postdose
  AUC (0-infinity) is the is the area under the plasma concentration-time curve from time zero to infinite time, calculated using the observed value of the last non-zero plasma concentration and will be evaluated when compared for 3 oral tablet formulations of seltorexant in fasted and semi-fasted conditions.
Relative Bioavailability of Seltorexant when Compared for 3 Oral Tablet Formulations of Seltorexant | Predose, 20 minutes (min), 30min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 20h (Day 1), 24h, 36h (Day 2), 48h (Day 3) postdose
  Relative bioavailability is the percentage of the administered dose that is systemically available, calculated as: (AUC [0-infinity] of test divided by AUC [0-infinity] of reference) multiplied by 100, where the reference treatment is a non-intravenous administration. Relative bioavailability will be evaluated when compared for 3 oral tablet formulations of seltorexant in fasted and semi-fasted conditions.

SECONDARY OUTCOMES:
Cmax when Compared Between Fasted and Semi-Fasted Conditions | Predose, 20 minutes (min), 30min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 20h (Day 1), 24h, 36h (Day 2), 48h (Day 3) postdose
  Cmax when compared between fasted and semi-fasted conditions will be evaluated for the 3 oral tablet formulations of seltorexant.
AUC (0-last) when Compared Between Fasted and Semi-Fasted Conditions | Predose, 20 minutes (min), 30min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 20h (Day 1), 24h, 36h (Day 2), 48h (Day 3) postdose
  AUC (0-last) when compared between fasted and semi-fasted conditions will be evaluated for the 3 oral tablet formulations of seltorexant.
AUC (0-infinity) when Compared Between Fasted and Semi-Fasted Conditions | Predose, 20 minutes (min), 30min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 20h (Day 1), 24h, 36h (Day 2), 48h (Day 3) postdose
  AUC (0-infinity) when compared between fasted and semi-fasted conditions will be evaluated for the 3 oral tablet formulations of seltorexant.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From Screening till End-of- Study (up to approximately 18 weeks)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRAHS, Salt Lake City, Utah, United States